CLINICAL TRIAL: NCT02400164
Title: A (M)Ulti-center, Prospective, (O)Pen Label, Uncontrolled Feasibility (S)Tudy to Assess the Safety and Effectiveness of an Automatic Low Flow (A)Scites (Alfa) Pump (I)n Patients With (C)Irrhosis and Refractory or Recurrent Ascites
Acronym: MOSAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-AAR-007
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Cirrhosis; Ascites
MeSH Terms: conditions — Fibrosis; Ascites

ARMS (1):
- alfapump system (Experimental): The Sequana Medical alfapump system is an implanted subcutaneous device with a rechargeable battery that moves ascitic fluid from the peritoneal cavity to the urinary bladder where it is eliminated by spontaneous diuresis.
  Interventions: Device: alfapump system

INTERVENTIONS:
Device: alfapump system — The Sequana Medical alfapump system is an implanted subcutaneous device with a rechargeable battery that moves ascitic fluid from the peritoneal cavity to the urinary bladder where it is eliminated by spontaneous diuresis.

SUMMARY:
The study is a multi-center, prospective, open label, uncontrolled feasibility study enrolling 30 patients with refractory or recurrent ascites and cirrhosis at up to 6 sites. Patients will be enrolled during a 6 month enrollment phase after which data will be collected for 12months with an initial analysis after 3 months. Extended follow-up for safety monitoring purposes will continue for the lifetime of the patient or until the device is explanted.

ELIGIBILITY:
Inclusion Criteria:

1. patients ≥ 21 years of age
2. recurrence of grade 3 ascites requiring paracentesis for symptom relief more frequently than once per month for a minimum of 2 of the prior 3 months
3. cirrhosis of any etiology
4. failure to respond to or intolerance to high dose diuretics
5. expected survival of greater than 3 months (MELD score ≤ 21)
6. screened for varices and on optimal management
7. diagnostic paracentesis with neutrophil count < 250 / µl within 24 hours of implantation
8. written informed consent
9. ability to comply with study procedures and ability to operate the device
10. women of childbearing potential should use adequate contraception

Exclusion Criteria:

1. more than 2 systemic or local infections, such as peritonitis, urinary tract infection, or abdominal skin infection within the last 6 months
2. presence of any current cancer
3. evidence of extensive ascites loculation
4. serum creatinine > 1.5 mg/dl
5. serum bilirubin > 5 mg/dl
6. eGFR < 30 ml/min/1.73m2 by MDRD (Modification of Diet in Renal Disease) method
7. gastrointestinal hemorrhage due to portal hypertension in the 2 weeks prior to inclusion in the study
8. hepatic encephalopathy > stage II in the two weeks prior to implant
9. presence of a patent TIPS or surgical portosystemic shunt
10. presence of Budd-Chiari syndrome
11. previous solid organ transplant
12. obstructive uropathy (bladder residual volume > 100ml (determined by catheterization or abdominal ultrasound) or any bladder anomaly which may contraindicate implantation of the alfapump, including recurrent urinary tract infections, vesicoureteral reflux, or history of urinary calculi)
13. International Prostate Symptom Score (I-PSS) ≥20
14. thrombocytopenia < 45,000 X106/l
15. patient undergoing therapeutic anticoagulation
16. recent (<4 months) intra-abdominal foreign body or abdominal surgery, diaphragmatic hernia, abdominal surgery, severe abdominal adhesions, surgically irreparable hernia, abdominal wall or skin infection, or severe malnutrition.
17. history (>6 months) of diaphragmatic hernia, history of bladder cancer, inflammatory or ischemic bowel disease, and frequent episodes of diverticulitis.
18. any non-liver disease with life expectancy < 1 year
19. patients eligible for TIPS (unless they have refused TIPS placement).
20. presence of any active implantable or body-worn devices that cannot be removed
21. pregnancy
22. patients being in another therapeutic clinical study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of serious adverse events related to the device and its implantation. | 12 months

SECONDARY OUTCOMES:
Assess the overall requirement for large volume paracentesis | 12 months
  Assess the overall requirement for large volume paracentesis by investigation of:
  * the number of large volume therapeutic paracentesis events and all paracentesis events
  * the annualized rate of large volume therapeutic paracentesis and of all paracentesis events
  * the cumulative volume of ascites removed through all paracentesis events
    • Assess the overall requirement for large volume paracentesis by investigation of:
  * the number of large volume therapeutic paracentesis events and all paracentesis events
  * the annualized rate of large volume therapeutic paracentesis and of all paracentesis events
  * the cumulative volume of ascites removed through all paracentesis events
Nutritional status | 12 months
  Nutritional status
  o evaluate changes in serum prealbumin
Evaluate patient quality of life | 12 months
  Evaluate patient quality of life
  * chronic liver disease questionnaire (CLDQ)
  * PLD questionnaire
  * ECOG performance status
Overall survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kamath, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (6):
- United States (5):
  - California Pacific Medical, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - Baylor University Healthcare System, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - VCU Medical Centre, Richmond, Virginia
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wong F, Bendel E, Sniderman K, Frederick T, Haskal ZJ, Sanyal A, Asrani SK, Capel J, Kamath PS. Improvement in Quality of Life and Decrease in Large-Volume Paracentesis Requirements With the Automated Low-Flow Ascites Pump. Liver Transpl. 2020 May;26(5):651-661. doi: 10.1002/lt.25724. Epub 2020 Mar 22. PMID 31999044